CLINICAL TRIAL: NCT02751632
Title: Staged Treatment in Early Psychosis (STEP): A Sequential Multistage Randomized Clinical Trial (SMART) of Interventions for Ultra High Risk (UHR) of Psychosis Patients.
Brief Title: The Staged Treatment in Early Psychosis Study
Acronym: STEP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orygen (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Davis (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2015.173; 1U01MH105258-01 (NIH)
Record Dates: First submitted 2016-04-12; First posted 2016-04-26 (Estimated); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Psychotic Disorders; Personality Disorders; Clinical High Risk
Keywords: Ultra High Risk of Psychosis; Prodrome; Clinical High Risk of Psychosis
MeSH Terms: conditions — Psychotic Disorders; Personality Disorders | interventions — Palliative Care; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (7):
- Step 1-Regular SPS Therapy (Experimental): Support and Problem Solving Therapy delivered to all study participants over a six-week period with a minimum of three sessions.
  Interventions: Behavioral: Support and Problem Solving Therapy
- Responders- Monthly SPS Therapy (Experimental): Participants are randomised to receive monthly Support and Problem Solving Therapy for up to 12 months.
  Interventions: Behavioral: Support and Problem Solving Therapy
- Responders- 3-monthly monitoring (Experimental): Participants are randomised to be monitored for risk every 3 months for up to 12 months.
  Interventions: Behavioral: 3-monthly monitoring
- Step 2- Regular SPS Therapy (Experimental): Participants are randomised to receive regular sessions of Support and Problem Solving Therapy, with a minimum of six sessions delivered over an 18-week period.
  Interventions: Behavioral: Support and Problem Solving Therapy
- Step 2- Regular CBCM (Experimental): Participants are randomised to receive regular sessions of Cognitive Behavioural Case Management, with a minimum of six sessions delivered over an 18-week period.
  Interventions: Behavioral: Cognitive Behavioural Case Management
- Step 3- Regular CBCM + Fluoxetine (Experimental): Participants are randomised to receive either Cognitive Behavioural Case Management plus an antidepressant medication for six months .
  Interventions: Behavioral: Cognitive Behavioural Case Management; Drug: Fluoxetine
- Step 3- Regular CBCM+ placebo (Placebo Comparator): Participants are randomised to receive Cognitive Behavioural Case Management plus placebo medication for six months.
  Interventions: Behavioral: Cognitive Behavioural Case Management; Drug: Placebo

INTERVENTIONS:
Behavioral: Support and Problem Solving Therapy — Support and Problem Solving Therapy involves providing participants with emotional support and helping them to resolve their problems in day-to-day life.
  Other Names: SPS
  Arms: Responders- Monthly SPS Therapy; Step 1-Regular SPS Therapy; Step 2- Regular SPS Therapy
Behavioral: Cognitive Behavioural Case Management — CBCM has a number of different elements including: strategies to help with stress management; therapy that targets thinking and behavioural patterns; practical assistance, as well as yoga and mindfulness.
  Other Names: CBCM
  Arms: Step 2- Regular CBCM; Step 3- Regular CBCM + Fluoxetine; Step 3- Regular CBCM+ placebo
Drug: Fluoxetine — Participants will commence on 1 capsule of fluoxetine 20 mg, to be taken in the morning. The medication can be increased to fluoxetine 40 mg daily if there has been a poor clinical response after the first 6 weeks of treatment.
  Other Names: Anti-depressant medication
  Arms: Step 3- Regular CBCM + Fluoxetine
Drug: Placebo — Participants will commence on 1 capsule of the placebo pill, to be taken in the morning. The medication can be increased to 2 placebo capsules if there has been a poor clinical response after the first 6 weeks of treatment.
  Other Names: Inactive Medicine
  Arms: Step 3- Regular CBCM+ placebo
Behavioral: 3-monthly monitoring — Study participants will be contacted on a 3-monthly basis by a study clinician who will be assessing the participant's risk.
  Arms: Responders- 3-monthly monitoring

SUMMARY:
A sequential multistage randomised clinical trial (SMART) to produce evidence to guide a step-wise clinical approach for the treatment of ultra high risk patients and reduction of risk for psychosis and other deleterious clinical and/or functional outcomes.

DETAILED DESCRIPTION:
The study treatment sequence involves three stages, which are referred to as steps:

Step 1- Support and Problem Solving (SPS)

All trial participants receive SPS treatment in Step 1. Step 1 involves attending weekly-fortnightly SPS sessions over a six week period and the Week 4 and 6 visits will also include an interview with research staff who will assess the symptoms and mental state of participants. These assessments will enable research staff to determine whether the therapy has been effective in improving the participant's symptoms.

Depending on how they respond to the six-week period of treatment in Step 1, participants are randomly assigned to a new treatment arm at the end of Step 1 as detailed below:

Participants who improve with the SPS treatment they receive during Step 1, will be randomised to either monthly SPS treatment for up to one year OR to three-monthly appointments (Month 3, 6, 9 and 12) to monitor their mental state.

Participants who do not improve with the SPS treatment they receive during Step 1 will be randomised to continue treatment in one of two groups in Step 2 as outlined below.

Step 2- Support and Problem Solving (SPS) OR Cognitive Behavioural Case Management (CBCM)

In Step 2, participants will receive either SPS OR Cognitive Behavioural Case Management for a period of 18 weeks. Participants will be interviewed at two time points across this step so that research staff can assess whether the therapy has helped improve their symptoms.

Participants who improve with the treatment they receive in Step 2 will be randomised to receive either monthly SPS for a further six months OR to three-monthly appointments (Month 9, 12) to monitor their mental state.

Participants who do not improve with the treatment they receive in Step 2 will be randomised to one of two treatment groups in Step 3 as outlined below.

Step 3 Cognitive Behavioural Case Management plus antidepressant medication OR Cognitive Behavioural Case Management plus placebo medication.

Participants assigned to one of the two treatment groups in Step 3 will receive the corresponding treatment over a six-month period. Both treatment groups will involve: regular CBCM sessions; regular review by a clinician, as well as the assigned medication.

Depending on which group participants are randomised to, they may either receive antidepressant medication OR placebo medication.

If a participant does not improve, or deteriorates by 12 weeks into Step 3, they will be given a choice to: continue with the treatment regime already assigned to them; increase the dosage of their medication, or start a new medication. Upon their choosing, the medication at this stage may either be an antipsychotic medication OR omega-3 fatty acids ('fish oil'), taken in addition to the other treatment components of this step.

The intervention aspect of this study covers a 12 month period. After completion of this intervention period, participants will also be invited to take part in two separate follow-up interviews with research staff, at both 18 months and 24 months.

US Pilot Study:

The University of California, Davis will oversee a pilot study for the implementation of the STEP model in the Early Diagnosis and Preventative Treatment (EDAPT) clinic at UC Davis in Sacramento, California. After giving informed consent, CHR patients and their families entering treatment in the EDAPT program will be offered participation in the staged intervention trial. CHR participants will be characterized with the Structured Interview for Prodromal Syndromes (SIPS) following standard procedures in the U.S. Similarly, defining risk based on 3 core syndromes that span analogous dimensions of symptom severity from attenuated to psychotic, a recent meta-analysis demonstrates that the SIPS reliably identifies youth at clinical high risk for psychosis at a rate comparable to the CAARMS, which is used in the main trial being conducted in the Orygen parent study. Thirty patients will be enrolled and followed through the protocol until 24 month follow up.The team will also harmonize CBT practice with the CBCM model used at Orygen. All outcome measures will parallel those used in the parent study at Orygen. UC Davis research staff will complete clinical and outcome assessments with CHR participants at study entry, 6, 12 and 24 months. Data analysis will also parallel those conducted in the parent study. However, the key measures will be acceptance and retention in the staged treatment.

US Focus Groups:

The University of California, San Francisco will design, conduct and analyze output from a series of focus groups to gather input from stakeholders regarding translation of STEP trial interventions to the US healthcare system. This will include identifying barriers and solutions to implementation of STEP trial interventions in the US context for CHR patients. Groups will include CA county mental health leadership, private insurance mental health leadership, mental health leadership at DHHS and the Center for Medicare/Medicaid Services, leadership from community-based organizations currently providing services for this population, consumers, and family members.

ELIGIBILITY:
INCLUSION CRITERIA

* Age 12 -25 years (inclusive) at entry.
* Ability to speak adequate English (for assessment purposes).
* Ability to provide informed consent.
* Meeting one or more Ultra High Risk for psychosis groups as defined below:

Group 1: Vulnerability Group

Family history of psychosis in first degree relative OR Schizotypal Personality Disorder (as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM) IV in identified patient

AND

Drop in Functioning:

Recency: Change in functioning occurred within last year Impact: Social and Occupational Functioning Assessment Scale (SOFAS) score at least 30% below previous level of functioning and sustained for at least one month.

OR

Sustained low functioning:

Recency: For the past 12 months or longer Impact: SOFAS score of 50 or less.

Group 2: Attenuated Psychotic Symptoms Group 2a) Subthreshold intensity:

Intensity: Global Rating Scale Score of 3-5 on Unusual Thought Content subscale, 3-5 on Non-Bizarre Ideas subscale, 3-4 on Perceptual Abnormalities subscale and/or 4-5 on Disorganised Speech subscales of the Comprehensive Assessment of At Risk Mental States (CAARMS).

Frequency: Frequency Scale Score of 3-6 on Unusual Thought Content, Non-Bizarre Ideas, Perceptual Abnormalities and/or Disorganised Speech subscales of the CAARMS

Duration: symptoms present for at least one week

Recency: symptoms present in past year

2b) Subthreshold frequency:

Intensity: Global Rating Scale Score of 6 on Unusual Thought Content subscale, 6 on Non-Bizarre Ideas subscale, 5-6 on Perceptual Abnormalities subscale and/or 6 on Disorganised Speech subscales of the CAARMS

Frequency: Frequency Scale Score of 3 on Unusual Thought Content, Non-Bizarre Ideas, Perceptual Abnormalities and/or Disorganised Speech subscales of the CAARMS

Recency: symptoms present in past year

Group 3: Brief Limited Intermittent Psychotic Symptoms Intensity: Global Rating Scale Score of 6 on Unusual Thought Content subscale, 6 on Non-Bizarre Ideas subscale, 5 or 6 on Perceptual Abnormalities subscale and/or 6 on Disorganised Speech subscales of the CAARMS

Frequency: Frequency Scale Score of 4-6 on Unusual Thought Content, Non-Bizarre Ideas, Perceptual Abnormalities and/or Disorganised Speech subscales

Duration: Symptoms present for less than one week and spontaneously remit on every occasion.

Recency: symptoms present in past year

EXCLUSION CRITERIA

* Past history of a psychotic episode of one week or longer, whether treated with antipsychotic medications or not.
* Attenuated psychotic symptoms only present during acute intoxication.
* Organic brain disease known to cause psychotic symptoms, e.g. temporal lobe epilepsy.
* Any metabolic, endocrine or other physical illness, e.g. thyroid disease, with known neuropsychiatric consequences.
* Diagnosis of a serious developmental disorder, e.g. Severe Autism Spectrum Disorder.
* Premorbid Intelligence Quotient (IQ) <70 and a documented history of developmental delay or intellectual disability.
* Current or previous SCID diagnosis of Bipolar I.

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 342 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Global Functioning Scale Score | 6 months from baseline (end of Step 2)
  To test the effect of a sequential treatment approach consisting of SPS/SPS and SPS/CBCM on functioning levels of UHR patients.

SECONDARY OUTCOMES:
Global Functioning Scale Score | 12 months from baseline (end of Step 3)
  To test the effect of a sequential treatment approach consisting of SPS, CBCM and antidepressant medication on functioning levels of UHR patients.
Comprehensive Assessment of At Risk Mental State score | 12 and 24 months from baseline
  To test the effect of a sequential treatment approach consisting of SPS, CBCM and antidepressant medication on transition to psychotic disorder.
Comprehensive Assessment of At Risk Mental State score | 1.5, 6, 12 and 24 months from baseline
  To test the effect of a sequential treatment approach on UHR status (maintenance versus remission).
Scale for Assessment of Negative Symptoms score | 1.5, 6, 12 and 24 months from baseline
  To test the effect of a sequential treatment approach in UHR patients on level of negative psychotic symptoms.
Comprehensive Assessment of At Risk Mental State score | During the first 12 months from baseline.
  To test relapse rates (to UHR+ status) in the relapse prevention/responder arm of the trial (SPS v monitoring).
Montgomery Asberg Depression Rating Scale score | 1.5, 6, 12 and 24 months from baseline
  To test the effect of a sequential treatment approach in UHR patients on level and depressive symptoms.
Comprehensive Assessment of At Risk Mental State score | 1.5, 6, 12 and 24 months from baseline
  To test the effect of a sequential treatment approach in UHR patients on level of positive psychotic symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McGorry, MD, PhD, Principal Investigator — Orygen Youth Research Centre
Locations (5):
- Australia (5):
  - Headspace, Craigieburn, Victoria
  - Headspace, Glenroy, Victoria
  - Orygen Youth Health Clinical Program, Melbourne, Victoria
  - Headspace, Sunshine, Victoria
  - Headspace, Werribee, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGorry PD, Mei C, Amminger GP, Yuen HP, Kerr M, Spark J, Wallis N, Polari A, Baird S, Buccilli K, Dempsey SA, Ferguson N, Formica M, Krcmar M, Quinn AL, Mebrahtu Y, Ruslins A, Street R, Wannan C, Dixon L, Carter C, Loewy R, Niendam TA, Shumway M, Nelson B. A Sequential Adaptive Intervention Strategy Targeting Remission and Functional Recovery in Young People at Ultrahigh Risk of Psychosis: The Staged Treatment in Early Psychosis (STEP) Sequential Multiple Assignment Randomized Trial. JAMA Psychiatry. 2023 Sep 1;80(9):875-885. doi: 10.1001/jamapsychiatry.2023.1947. PMID 37378974